CLINICAL TRIAL: NCT02848924
Title: Current Incidence and Treatments Performed of Fractures of the Acetabulum and Pelvis in France in 2013
Acronym: ACETABULUM
Status: Completed | Type: Observational
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: ACETABULUM
Record Dates: First submitted 2016-07-21; First posted 2016-07-29 (Estimated); Last update posted 2016-07-29 (Estimated); Status verified 2016-07

CONDITIONS: Acetabulum; Fractures
Keywords: prevalence; surgery; Treatments
MeSH Terms: conditions — Fractures, Bone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: No intervention

SUMMARY:
Fractures of the acetabulum and pelvis are serious injuries to vital prognostic can play in cases of severe bleeding. In all cases the functional is a major issue with a potential reach of walking ability and maintaining the seated and standing positions. The treatment of such lesions requires management to a specialist, or the ability to use such centers for advice or transferring patients. This organization was recommended after the symposium of the French Society of Orthopedic Surgery (SOFCOT) in 2009. With the aging population, the incidence and clinical features of these fractures have evolved to worsening the functional prognosis. Club Basin acetabulum, body SOFCOT, wants to achieve an observational study assessing needs and practices at national and regional level. The long-term objective is to propose a regional organization of care of these patients in order to reduce morbidity and mortality associated.

DETAILED DESCRIPTION:
Fractures of the acetabulum and pelvis are serious injuries to vital prognostic can play in cases of severe bleeding. In all cases the functional is a major issue with a potential reach of walking ability and maintaining the seated and standing positions. The treatment of such lesions requires management to a specialist, or the ability to use such centers for advice or transferring patients. This organization was recommended after the symposium of the French Society of Orthopedic Surgery (SOFCOT) in 2009. With the aging population, the incidence and clinical features of these fractures have evolved to worsening the functional prognosis. Club Basin acetabulum, body SOFCOT, wants to achieve an observational study assessing needs and practices at national and regional level. The long-term objective is to propose a regional organization of care of these patients in order to reduce morbidity and mortality associated.

FORMAT OF RESEARCH retrospective observational study of SNIIRAM data on hospitalizations for broken pelvis and acetabulum (CCAM codes S32.40 / S32.41 / S32.30 / S32.31 / S32.10 / S32.11 / S32.50 / S32 .51 / S32.70 / S32.71 / S32.80 / S32.81), with collection of the following data:

* Patient demographics: age, sex, comorbidities (DRG coding), place of residence.
* Length of hospital stay
* Treatment undertaken: CCAM coding during hospitalization
* Mortality at 30 days and 1 year.

ELIGIBILITY:
Inclusion Criteria:

* All patients

Exclusion Criteria:

* No exclusion criteria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients hospitalized for broken pelvis and acetabulum in France
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2015-01; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Assessment of hospital stay length from medical file | Day 1 after hospitalization
Assesment of change of mortality | Day 30 and 1 year after hospitalization
  Assesment of change of mortality in this point time using a phone call.

CONTACTS AND LOCATIONS:
Overall Officials: JOUFFROY Pommes, MD, Principal Investigator — Fondation Hôpital Saint-Joseph
Locations (1):
- Groupe Hospitalier Paris Saint Joseph, Paris, Île-de-France Region, France